CLINICAL TRIAL: NCT06906575
Title: "Walking Together with Love": a Comprehensive Intervention Targeting Body Image, Psychological Flexibility, and Dyadic Coping for Sexual and Relationship Distress Among Cancer Patients and Their Partners
Brief Title: "Walking Together with Love": a Couples-Based Intervention for Sexual and Relationship Distress in Cancer Patients
Acronym: WTL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yanfei Jin (Other)
Responsible Party: Sponsor-Investigator, Yanfei Jin, Nanjing Medical University, Central South University
Organization: Central South University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-749; 2024-749 (Registry Identifier: Nanjing Medical University Ethics Committee)
Record Dates: First submitted 2025-03-24; First posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Sexual Dysfunction, Psychological; Relationship Distress; Cancer
MeSH Terms: conditions — Sexual Dysfunctions, Psychological; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Walking Together with Love (Experimental)
  Interventions: Behavioral: A Comprehensive Intervention to Improve Sexual and Relationship Well-being for Cancer Patients and Their Partners

INTERVENTIONS:
Behavioral: A Comprehensive Intervention to Improve Sexual and Relationship Well-being for Cancer Patients and Their Partners — This intervention targets three core areas:
  Body Image Improvement - Supports patients in understanding and accepting physical changes resulting from cancer treatments, fostering positive attitudes toward body image and self-esteem.
  Psychological Flexibility Enhancement - Utilizes ACT-based strategies to help participants acknowledge and adaptively manage difficult emotions, thoughts, and experiences related to cancer diagnosis and treatment.
  Dyadic Coping Skill Training - Provides structured skill-building exercises to strengthen mutual support mechanisms, enhance effective partner communication, and promote collaborative problem-solving when facing cancer-related stressors.
  The intervention consists of six weekly sessions (90-120 minutes each), delivered in a hybrid format (virtual and in-person) to maximize accessibility. Each session integrates psychoeducational presentations, facilitated discussions, guided experiential exercises.

SUMMARY:
Cancer diagnosis and treatment often result in significant changes in body appearance, sexual functioning, and relationship quality, leading to distress for both patients and their partners. To address these challenges, a comprehensive intervention program called "Walking Together with Love" (WTL) has been developed.

This intervention focuses on three key areas: improving body image (supporting patients in accepting physical changes after cancer treatment), enhancing psychological flexibility (enabling patients and partners to openly and positively manage difficult experiences), and strengthening dyadic coping skills (promoting effective communication and emotional support between partners). The primary aim of this intervention is to reduce sexual and relationship distress among cancer patients and their partners.

WTL is a six-week program consisting of weekly 90- to 120-minute sessions delivered in a hybrid format (both online and offline). Sessions incorporate psychoeducational presentations, group discussions, professional guidance, and structured home assignments. Both patients and their partners participate together, collaboratively working toward improving relationship quality and overall well-being.

Cancer patients, their partners, and healthcare providers are encouraged to learn more about this research project and explore its potential benefits in improving quality of life for couples affected by cancer.

DETAILED DESCRIPTION:
Cancer diagnosis and treatment frequently lead to multiple physical, psychological, and interpersonal challenges. Among these, disruptions in body image, sexual functioning, and relationship dynamics are particularly common and distressing for both patients and their intimate partners. Existing evidence suggests that difficulties in accepting body changes, reduced psychological flexibility, and inadequate dyadic coping strategies significantly contribute to sexual and relationship distress among couples facing cancer.

To address these unmet needs, a couples-based intervention called "Walking Together with Love" (WTL) has been developed. Grounded in cognitive behavioral therapy (CBT), acceptance and commitment therapy (ACT), and dyadic coping theory, this intervention integrates three core therapeutic components:

Body Image Improvement:

Supports cancer patients and their partners in understanding and accepting physical changes resulting from cancer treatments.

Fosters positive attitudes toward body image and self-esteem.

Psychological Flexibility Enhancement:

Utilizes ACT-based strategies to improve participants' ability to acknowledge and adaptively manage difficult emotions, thoughts, and experiences related to cancer diagnosis and treatment.

Dyadic Coping Skill Training:

Provides systematic skill-building exercises designed to strengthen mutual support mechanisms, enhance effective communication, and promote collaborative problem-solving when facing cancer-related stressors.

The WTL intervention is delivered in a structured, interactive, and collaborative manner, specifically designed to support both patients and their partners.

Program Duration and Format:

A six-week structured intervention program, with weekly sessions lasting approximately 90-120 minutes.

Sessions are delivered in a hybrid format (virtual and in-person) to maximize accessibility and convenience.

Session Content and Methods:

Each session incorporates psychoeducational presentations, guided discussions, experiential exercises, and structured home assignments.

Core areas covered include managing body image concerns, cultivating psychological flexibility, enhancing intimacy and communication skills, and reinforcing collaborative coping strategies.

Participant Involvement:

Both cancer patients and their intimate partners actively engage in all sessions, participating in therapeutic tasks and home assignments.

This collaborative approach fosters mutual understanding, emotional closeness, and relationship resilience.

Evaluation and Outcome Measures:

To assess the effectiveness of the intervention, multiple time-point assessments will be conducted (pre-intervention baseline, post-intervention, and follow-up assessments).

Outcome measures include sexual and relationship distress, body image acceptance, psychological flexibility, relationship quality, and overall well-being, assessed using validated psychometric instruments.

The primary goal of the WTL intervention is to provide a practical, evidence-based, and scalable approach to alleviating sexual and relationship distress among cancer patients and their intimate partners. By addressing psychological and relational challenges, this intervention aims to enhance quality of life and psychosocial adjustment to cancer.

ELIGIBILITY:
Inclusion Criteria:

Diagnosed with cancer, with a duration of at least 3 months after surgery; Aged 18-49 and married; were able to complete the questionnaire independently; were willing to participate.

Exclusion Criteria: cognitive or psychiatric impairments and suffering from severe heart, liver, kidney, and other serious complications.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-10-26 (Estimated); Study Completion 2025-10-26 (Estimated)

PRIMARY OUTCOMES:
Sexual and Relationship Distress | 3 months after intervention
  The Sexual and Relationship Distress Scale (SaRDS) is used to measured the Sexual and Relationship Distress .The SaRDS is a 30-item, 14-factor patient-reported outcome measure of individual and relationship distress within the context of sexual dysfunction14. All items are rated on a 7-point Likert scale ("not at all true" to "completely true"). The total scores range from 0 to 180 and reflect the standard of individual and relationship distress within the context of sexual dysfunction, with high values indicating more distress. In the original version of the study, the SaRDS showed good psychometric properties, and the subsequent studies also reported the strong internal consistency of the SaRDS (Cronbach alpha = .95 for the total score with individual sub-scales ranging from .70-.96).
Relationship Satisfaction | 3 months after intervention
  The Couples Satisfaction Index (CSI-16) is a validated measure of relationship satisfaction, assessing perceived intimacy, emotional closeness, and overall satisfaction within the relationship. Higher scores indicate greater relationship satisfaction.

SECONDARY OUTCOMES:
Body Image | 3 months after intervention
  The Body Image Scale (BIS) will be used to assess body image concerns among cancer patients. The BIS is a validated 10-item self-report questionnaire designed to evaluate body image distress, self-consciousness, and changes in body perception following cancer treatment. Higher scores indicate greater body image disturbance.
Psychological Flexibility | 3 months after intervention
  Measurement Tool: The Acceptance and Action Questionnaire-II (AAQ-II) will be used to assess psychological flexibility. The AAQ-II is a validated 7-item self-report measure that evaluates experiential avoidance and the ability to accept thoughts and emotions while engaging in values-based actions. Higher scores indicate greater psychological inflexibility, while lower scores reflect higher psychological flexibility.
Dyadic Coping | 3 months after intervention
  Measurement Tool: The Dyadic Coping Inventory (DCI) will be used to assess dyadic coping strategies among cancer patients and their partners. The DCI is a validated self-report questionnaire that evaluates how partners support each other in managing stress, communicate emotions, and engage in joint coping efforts. Higher scores indicate more effective dyadic coping and greater relationship resilience.

IPD SHARING:
Plan to Share IPD: No